CLINICAL TRIAL: NCT06414694
Title: Inpatient Penicillin Delabeling for Low-Risk Patients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-09373-FB
Record Dates: First submitted 2024-04-25; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Penicillin; Drug Allergy
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Direct Challenge (Experimental): Patients who met enrollment criteria proceed to direct oral challenge with penicillin with one hour observation, 48 hour phone call, six month follow-up.
  Interventions: Procedure: Direct Oral Challenge

INTERVENTIONS:
Procedure: Direct Oral Challenge — Direct oral challenge to penicillin at a goal dose of 45 mg/kg given in a 10%/90% dose

SUMMARY:
This study seeks to enroll patients admitted to a children's hospital with identified penicillin allergy. A screening checklist is performed to identify patients with very low or low risk histories of penicillin allergy to offer direct oral challenges to the antibiotic class to de-label patient's with drug allergies.

DETAILED DESCRIPTION:
This is a pilot study looking to utilize a novel criterion to identify low risk penicillin allergies for patients admitted to a children's hospital to evaluate safety and efficacy of direct oral challenges to patients with very low or low risk histories as identified in novel criterion.

ELIGIBILITY:
Inclusion Criteria:

* Patients >2 years
* Patients identified via EMR as having a penicillin, amoxicillin, amoxicillin/clavulanic acid allergy

Exclusion Criteria:

* Female patients aged >8 years of age
* Patients with hemodynamic instability
* Patients identified with moderate or high risk histories per protocol
* Patients currently taking oral antihistamines in 48 hours prior to direct challenge
* Patients currently taking oral steroids in 48 hours prior to direct challenge
* Patients currently receiving medications for nausea, shortness of breath,

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Direct Oral Challenge | 2 hours
  Pass or Failure of direct oral challenge

SECONDARY OUTCOMES:
Follow-up at 48 | 48 hours
  Follow-up phone call to assess adverse reaction by 48 hours. Data to be collected by screening questionnaire to assess for reactions such as fever, rash, manufacturer labeled adverse side effects.
Follow-up at 6 months | 6 months
  Follow-up phone call to assess subsequent tolerance or reaction of penicillin based antibiotic if prescribed in this time period. Data to be collected by screening questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No